CLINICAL TRIAL: NCT06241586
Title: A Novel Surgical Strategy to Reduce Major Complications in Patients With Necrotizing Pancreatitis: A Retrospective Cohort Study
Brief Title: A Novel Surgical Strategy to Reduce Major Complications in Patients With Necrotizing Pancreatitis
Status: Completed | Type: Observational
Sponsor: Tianjin Nankai Hospital (Other)
Responsible Party: Principal Investigator, Yang Yang, Resident physicians, Tianjin Nankai Hospital
Other Study IDs: TianjinNH
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the early period group: Patients admitted before January 2021 received the hybrid strategy of traditional and novel surgical strategies.
  Interventions: Procedure: The novel PMMI surgical strategy; Procedure: The conventional step-up strategy
- the late period group: Patients admitted during and after January 2021 received the complete novel PMMI surgical strategy.
  Interventions: Procedure: The novel PMMI surgical strategy

INTERVENTIONS:
Procedure: The novel PMMI surgical strategy — Immediate drainagewas advocated within 24 hours once necrosis was diagnosed. During the treatment course, a hybrid approach was available by flexibly switching interventions. Open surgery was only applied when patients required emergency surgery.
  The minimally invasive surgery was selected based on the size, location, and maturity of the necrotic area and stepwise response to intervention. Repeated peritoneal purification was performed until the infected or devitalized tissue was controlled. Patients were subsequently discharged with a drainage catheter and readmitted at 7- to 10-day intervals to receive repeated planned surgery without postoperative irrigation. Patients received a whole-course assessment for individual patients at 7-day predetermined intervals.
Procedure: The conventional step-up strategy — Interventions were postponed until 4 weeks after the onset of pancreatitis in line with international guidelines unless the patient showed evidence of progressive clinical deterioration despite the use of maximal supportive care. Patients underwent CT-guided percutaneous catheter drainage as the first step. Treatment response was evaluated after 3 days. If drainage was clinically unsuccessful, a VARD procedure was performed. Similarly, open surgery, which was described by Beger et al., was performed if the VARD procedure failed. Postoperative continuous lavage is performed as a routine procedure.
  Groups: the early period group

SUMMARY:
The goal of this observational study is to compare patient outcomes between the groups of patients admitted before and after the full implementation of the novel surgical strategy in patients with necrotizing pancreatitis. The main question it aims to answer are:

• the efficacy and safety of the novel surgical strategy To assess the efficacy and safety of the novel surgical strategy, all included patients were divided into two groups according to the timing of receiving treatment: 1) the early period group: patients admitted before January 2021 received the hybrid strategy of traditional and novel surgical strategies; and 2) the late period group: patients admitted during and after January 2021 received the complete novel surgical strategy.

ELIGIBILITY:
Inclusion Criteria:

Consecutive patients older than 18 years with necrotizing pancreatitis were included.

Exclusion Criteria:

Patients who met one or more of the following criteria were excluded: (1) had a past medical history of acute pancreatitis; (2) had drainage or surgery for pancreatic necrosis in other hospitals before admission to our institute; and (3) did not complete the treatment strategy owing to nonmedical reasons.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We conducted a retrospective, before-after, single-center study from January 2019 to September 2022 at the Department of Surgery, Tianjin Nankai Hospital. Consecutive patients older than 18 years with necrotizing pancreatitis were included.
Sampling Method: Non-Probability Sample
Enrollment: 271 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
major complications | 90-day follow up

SECONDARY OUTCOMES:
mortality | 90-day follow up
Admission of ICU | up to 90-days
Length of hospital stay | up to 90-days
individual major complications | 90-day follow up
  The overall complications included procedure-related complications (intra-abdominal and gastrointestinal bleeding, pancreatic fistulas, and gastrointestinal perforation) and nonspecific complications (systemic inflammatory response syndrome, abdominal compartment syndrome, and new-onset renal, respiratory and circulatory failure).

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin NanKai Hospital, Tianjin, None Selected, China

IPD SHARING:
Plan to Share IPD: No